CLINICAL TRIAL: NCT04796753
Title: Detection of Neuromuscular Deficits in Movement Pattern in Uninjured Federated Youth Basketball Players: a Cross-sectional Study
Brief Title: Detection of Neuromuscular Deficits in Uninjured Youth Basketball Players
Acronym: DPL
Status: Completed | Type: Observational
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, CRISTINA ADILLÓN, Associate Professor, University Rovira i Virgili
Other Study IDs: 123/2018
Record Dates: First submitted 2021-03-03; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Injury;Sports; Biomechanical Lesions; Musculoskeletal Injury
Keywords: Basketball; Physical Therapy; Youth athletes
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth basketball players who belonged to basketball developmental teams (U12, U14,U16,U17).: All participants completed the same ten-minute neuromuscular warm-up consisting of the following exercises: joint mobility exercises, dynamic stretching exercises, jumps, multidirectional displacements and changes of direction. Following, subjects were allowed three practice trials for each test. Consistent feedback was provided throughout to ensure proper technique. The performance of each test was recorded using two cameras (Iphone XS, Apple). To allow visible tracking of the different joints, participants were required to wear shorts with the hem at approximately mid-thigh. When scoring performance, each test was viewed in both planes (sagittal and frontal views).
  Interventions: Other: Basketball Injury Defense

INTERVENTIONS:
Other: Basketball Injury Defense — To establish a specific evaluation protocol for youth basketball players.

SUMMARY:
Basketball is an impact, coordination-opposition sport with continuous contact among players and it is considered a sport of medium-high injury incidence. Players are force to have a physical condition appropriate to their practice and the demand to which they must respond due to the intensity of the efforts this sport requires. In order to achieve this, it is necessary to establish an evaluation protocol that allows the detection of functional deficiencies, to guide and conduct in a specific and early way every moment of players' health and growth.

The purpose of this study is to evaluate and detect federated youth basketball players' (U12 - U17) neuromuscular deficiencies in mobility, stability and landing technique in static and dynamic situations to simulate all the most important actions of basketball demands.

DETAILED DESCRIPTION:
It is intended that the specific detection and individualized approach to neuromuscular deficiencies will decrease the prevalence of injuries and accidents and therefore, the performance of training basketball players will be improved. The purpose of this study was to evaluate and detect federated youth basketball players' (under 12 years until under 17 years) neuromuscular deficits in mobility, stability and landing technique in static and dynamic situations similar to simulate the most important actions of basketball demands.

This cross-sectional study was conducted from October 2018 to May 2019. A total of 778 basketball players were selected for the present study. In order to evaluate this specific tests and trials will be carried out on different teams from various clubs in the categories from under 12 years (U12) to under 17 (U17), both male and female. The evaluations will consist of a static physical measures and a dynamic one. These will be conducted throughout the season. Inclusion criteria were: age > 12 years and <18 years at testing, and to be actively competing during the study. Subjects were excluded if they had suffered any injury in lower limbs before the screening; presented any injury (overuse or acute) at the time of testing or if they suffered any oncological, psychological and/or psychiatric illnesses, or if they did not attend on the day of the assessment. The main outcomes were ankle joint dorsiflexion was analyzed with Weight-bearing Dorsiflexion Test; monopodial ankle stability was analyzed with Single Leg Balance Test. Dynamic lower extremity valgus was analyzed with Single Leg Squat Test, Modified Tuck Jump Test, Single Leg Squat Test and Hurdle Step Test were used to evaluate also Lumbopelvic stability and dynamic postural control. Neuromuscular deficits during continuous tuck jumps, landing technique flaws and Plyometric Technique were analyzed with Modified Tuck Jump Test. All these tests are scientifically validated for this purpose. All players were familiar with the procedures of all test before. Testing was performed in the same day, in the same order, at the same time of the day (18:00-20:00).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years and <18 years at testing.
* To be actively competing during the study.

Exclusion Criteria:

* Had suffered any injury in lower limbs before the screening.
* Presented any injury (overuse or acute) at the time of testing.
* Psychological or psychiatric diseases diagnosed.
* Oncological diseases diagnosed.
* Did not attend on the day of the assessment.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants were recruited through the Catalan Basketball Federation, and the study was carried out in the sports facilities of each club.
Sampling Method: Probability Sample
Enrollment: 575 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Ankle joint dorsiflexion | Through study completion, an average of 1 year
  Weight-bearing dorsiflexion test. Ankle dorsiflexion was evaluated through the LegMotion system (LegMotion, your Motion®, Albacete, Spain). Each player started with their hands on their hips, and put the assigned foot on the middle of the longitudinal line just behind the transversal line on the platform. The alternate foot was positioned off the platform with toes at the edge of the platform. Each trial consisted of flexing the ankle as much as possible without raising the heel of the assessed ankle trying to touch a marker, situated just behind the patella, with their knee. The distance achieved was recorded in centimeters. Three trials were allowed with each ankle (i.e., left and right) with 10 seconds of passive recovery between trials. The third value in each ankle was used in subsequent analysis of weight-bearing dorsiflexion.
Ankle stability | Through study completion, an average of 1 year
  Single Leg Balance Test. It was considered stable if the foot remained in neutral position during movement. However, if excessive pronation of the foot was evident during movement or external rotation of the leg/foot it was scored as unstable.
Dynamic lower extremity valgus | Through study completion, an average of 1 year
  Single Leg Squat Test. An aligned knee-ankle position was considered when the patella was aligned with the second toe. Five consecutive attempts were performed with each limb, and the correct alignment between the knee and the second toe in loading was assessed to analyze an excess of knee valgus.
Lumbopelvic stability | Through study completion, an average of 1 year
  Single Leg Squat Test. It was considered stable if there was minimal movement in all three planes and the sacroiliac joints were aligned. On the other hand, it was considered unstable if the sacroiliac joints were not aligned in the frontal plane or if there was evidence of anteroposterior tilt or rotation in the sagittal plane as well as anterior trunk flexion or increased lumbar lordosis.
Dynamic postural control | Through study completion, an average of 1 year
  Hurdle Step Test. For this purpose, the deviation of the trunk with respect to the center of gravity was observed. A smaller displacement or deviation implied a better postural stability.
Neuromuscular deficits during continuous tuck jumps | Through study completion, an average of 1 year
  Modified Tuck Jump Test. Lower extremity valgus at landing, Thighs do not reach parallel (peak of jump), Thighs not equal side-to-side during flight
Landing technique flaws | Through study completion, an average of 1 year
  Modified Tuck Jump Test. Foot placement not shoulder width apart, Foot placement not parallel (front to back), Foot contact timing not equal (Asymmetrical landing), Excessive landing contact noise.
Plyometric Technique | Through study completion, an average of 1 year
  Modified Tuck Jump Test. Pause between jumps, Technique declines prior 10 seconds, Does not land in same foot print (Consistent point of landing)

SECONDARY OUTCOMES:
Age | Through study completion, an average of 1 year
  Years
Age categories | Through study completion, an average of 1 year
  Under 12, Under 14, Under 16 or Under 17
Body Mass Index (BMI) | Through study completion, an average of 1 year
  kg/m2
Generalized hipermobility | Through study completion, an average of 1 year
  The presence of hypermobile confirmed by Beighton's criteria. Considering hypermobile as those who obtained a score of > 7 points out of a total of 9 points
Gender | Through study completion, an average of 1 year
  Female or male
Weight | Through study completion, an average of 1 year
  Kilograms
Height | Through study completion, an average of 1 year
  Centimeters
Wingspan | Through study completion, an average of 1 year
  Centimeters
Lower limb dominance | Through study completion, an average of 1 year
  Dominant leg / non dominant leg

CONTACTS AND LOCATIONS:
Locations (1):
- Federación Catalana de Baloncesto, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drakos MC, Domb B, Starkey C, Callahan L, Allen AA. Injury in the national basketball association: a 17-year overview. Sports Health. 2010 Jul;2(4):284-90. doi: 10.1177/1941738109357303. PMID 23015949
- [Background] Hootman JM, Dick R, Agel J. Epidemiology of collegiate injuries for 15 sports: summary and recommendations for injury prevention initiatives. J Athl Train. 2007 Apr-Jun;42(2):311-9. PMID 17710181
- [Background] Rodas G, Bove T, Caparros T, Langohr K, Medina D, Hamilton B, Sugimoto D, Casals M. Ankle Sprain Versus Muscle Strain Injury in Professional Men's Basketball: A 9-Year Prospective Follow-up Study. Orthop J Sports Med. 2019 Jun 21;7(6):2325967119849035. doi: 10.1177/2325967119849035. eCollection 2019 Jun. PMID 31259184
- [Background] Cherni Y, Jlid MC, Mehrez H, Shephard RJ, Paillard T, Chelly MS, Hermassi S. Eight Weeks of Plyometric Training Improves Ability to Change Direction and Dynamic Postural Control in Female Basketball Players. Front Physiol. 2019 Jun 13;10:726. doi: 10.3389/fphys.2019.00726. eCollection 2019. PMID 31263427
- [Background] Taylor JB, Wright AA, Dischiavi SL, Townsend MA, Marmon AR. Activity Demands During Multi-Directional Team Sports: A Systematic Review. Sports Med. 2017 Dec;47(12):2533-2551. doi: 10.1007/s40279-017-0772-5. PMID 28801751
- [Background] Zuckerman SL, Wegner AM, Roos KG, Djoko A, Dompier TP, Kerr ZY. Injuries sustained in National Collegiate Athletic Association men's and women's basketball, 2009/2010-2014/2015. Br J Sports Med. 2018 Feb;52(4):261-268. doi: 10.1136/bjsports-2016-096005. Epub 2016 Jun 30. PMID 27364907
- [Background] Andreoli CV, Chiaramonti BC, Buriel E, Pochini AC, Ejnisman B, Cohen M. Epidemiology of sports injuries in basketball: integrative systematic review. BMJ Open Sport Exerc Med. 2018 Dec 27;4(1):e000468. doi: 10.1136/bmjsem-2018-000468. eCollection 2018. PMID 30687514
- [Background] Pasanen K, Ekola T, Vasankari T, Kannus P, Heinonen A, Kujala UM, Parkkari J. High ankle injury rate in adolescent basketball: A 3-year prospective follow-up study. Scand J Med Sci Sports. 2017 Jun;27(6):643-649. doi: 10.1111/sms.12818. Epub 2016 Dec 29. PMID 28033652
- [Background] Leppanen M, Pasanen K, Kannus P, Vasankari T, Kujala UM, Heinonen A, Parkkari J. Epidemiology of Overuse Injuries in Youth Team Sports: A 3-year Prospective Study. Int J Sports Med. 2017 Oct;38(11):847-856. doi: 10.1055/s-0043-114864. Epub 2017 Sep 11. PMID 28895620
- [Background] Emery CA. Risk factors for injury in child and adolescent sport: a systematic review of the literature. Clin J Sport Med. 2003 Jul;13(4):256-68. doi: 10.1097/00042752-200307000-00011. PMID 12855930
- [Background] Agresta C, Church C, Henley J, Duer T, O'Brien K. Single-Leg Squat Performance in Active Adolescents Aged 8-17 Years. J Strength Cond Res. 2017 May;31(5):1187-1191. doi: 10.1519/JSC.0000000000001617. PMID 27575249
- [Background] Moseid CH, Myklebust G, Slaastuen MK, Bar-Yaacov JB, Kristiansen AH, Fagerland MW, Bahr R. The association between physical fitness level and number and severity of injury and illness in youth elite athletes. Scand J Med Sci Sports. 2019 Nov;29(11):1736-1748. doi: 10.1111/sms.13498. Epub 2019 Jul 1. PMID 31206837
- [Background] Monfort SM, Comstock RD, Collins CL, Onate JA, Best TM, Chaudhari AM. Association between ball-handling versus defending actions and acute noncontact lower extremity injuries in high school basketball and soccer. Am J Sports Med. 2015 Apr;43(4):802-7. doi: 10.1177/0363546514564541. Epub 2015 Jan 16. PMID 25596616
- [Background] Bahr R, Krosshaug T. Understanding injury mechanisms: a key component of preventing injuries in sport. Br J Sports Med. 2005 Jun;39(6):324-9. doi: 10.1136/bjsm.2005.018341. PMID 15911600
- [Background] Clifton DR, Hertel J, Onate JA, Currie DW, Pierpoint LA, Wasserman EB, Knowles SB, Dompier TP, Comstock RD, Marshall SW, Kerr ZY. The First Decade of Web-Based Sports Injury Surveillance: Descriptive Epidemiology of Injuries in US High School Girls' Basketball (2005-2006 Through 2013-2014) and National Collegiate Athletic Association Women's Basketball (2004-2005 Through 2013-2014). J Athl Train. 2018 Nov;53(11):1037-1048. doi: 10.4085/1062-6050-150-17. PMID 30715913
- [Background] Clifton DR, Onate JA, Hertel J, Pierpoint LA, Currie DW, Wasserman EB, Knowles SB, Dompier TP, Marshall SW, Comstock RD, Kerr ZY. The First Decade of Web-Based Sports Injury Surveillance: Descriptive Epidemiology of Injuries in US High School Boys' Basketball (2005-2006 Through 2013-2014) and National Collegiate Athletic Association Men's Basketball (2004-2005 Through 2013-2014). J Athl Train. 2018 Nov;53(11):1025-1036. doi: 10.4085/1062-6050-148-17. PMID 30715912
- [Background] Bond CW, Dorman JC, Odney TO, Roggenbuck SJ, Young SW, Munce TA. Evaluation of the Functional Movement Screen and a Novel Basketball Mobility Test as an Injury Prediction Tool for Collegiate Basketball Players. J Strength Cond Res. 2019 Jun;33(6):1589-1600. doi: 10.1519/JSC.0000000000001944. PMID 28426513
- [Background] Cook G, Burton L, Hoogenboom BJ, Voight M. Functional movement screening: the use of fundamental movements as an assessment of function - part 1. Int J Sports Phys Ther. 2014 May;9(3):396-409. PMID 24944860
- [Background] Tummala SV, Hartigan DE, Makovicka JL, Patel KA, Chhabra A. 10-Year Epidemiology of Ankle Injuries in Men's and Women's Collegiate Basketball. Orthop J Sports Med. 2018 Nov 5;6(11):2325967118805400. doi: 10.1177/2325967118805400. eCollection 2018 Nov. PMID 30480010
- [Background] Calatayud J, Martin F, Gargallo P, Garcia-Redondo J, Colado JC, Marin PJ. The validity and reliability of a new instrumented device for measuring ankle dorsiflexion range of motion. Int J Sports Phys Ther. 2015 Apr;10(2):197-202. PMID 25883868
- [Background] Bennell KL, Talbot RC, Wajswelner H, Techovanich W, Kelly DH, Hall AJ. Intra-rater and inter-rater reliability of a weight-bearing lunge measure of ankle dorsiflexion. Aust J Physiother. 1998;44(3):175-180. doi: 10.1016/s0004-9514(14)60377-9. PMID 11676731
- [Background] Trojian TH, McKeag DB. Single leg balance test to identify risk of ankle sprains. Br J Sports Med. 2006 Jul;40(7):610-3; discussion 613. doi: 10.1136/bjsm.2005.024356. Epub 2006 May 10. PMID 16687483
- [Background] Ugalde V, Brockman C, Bailowitz Z, Pollard CD. Single leg squat test and its relationship to dynamic knee valgus and injury risk screening. PM R. 2015 Mar;7(3):229-35; quiz 235. doi: 10.1016/j.pmrj.2014.08.361. Epub 2014 Aug 8. PMID 25111946
- [Background] Crossley KM, Zhang WJ, Schache AG, Bryant A, Cowan SM. Performance on the single-leg squat task indicates hip abductor muscle function. Am J Sports Med. 2011 Apr;39(4):866-73. doi: 10.1177/0363546510395456. Epub 2011 Feb 18. PMID 21335344
- [Background] Whatman C, Hume P, Hing W. The reliability and validity of physiotherapist visual rating of dynamic pelvis and knee alignment in young athletes. Phys Ther Sport. 2013 Aug;14(3):168-74. doi: 10.1016/j.ptsp.2012.07.001. Epub 2012 Oct 26. PMID 23107340
- [Background] Ageberg E, Bennell KL, Hunt MA, Simic M, Roos EM, Creaby MW. Validity and inter-rater reliability of medio-lateral knee motion observed during a single-limb mini squat. BMC Musculoskelet Disord. 2010 Nov 16;11:265. doi: 10.1186/1471-2474-11-265. PMID 21080945
- [Background] Cook G, Burton L, Hoogenboom B. Pre-participation screening: the use of fundamental movements as an assessment of function - part 1. N Am J Sports Phys Ther. 2006 May;1(2):62-72. PMID 21522216
- [Background] Fort-Vanmeerhaeghe A, Montalvo AM, Lloyd RS, Read P, Myer GD. Intra- and Inter-Rater Reliability of the Modified Tuck Jump Assessment. J Sports Sci Med. 2017 Mar 1;16(1):117-124. eCollection 2017 Mar. PMID 28344460
- [Background] Herrington L, Myer GD, Munro A. Intra and inter-tester reliability of the tuck jump assessment. Phys Ther Sport. 2013 Aug;14(3):152-5. doi: 10.1016/j.ptsp.2012.05.005. Epub 2012 Oct 16. PMID 23084318
- [Background] Smits-Engelsman B, Klerks M, Kirby A. Beighton score: a valid measure for generalized hypermobility in children. J Pediatr. 2011 Jan;158(1):119-23, 123.e1-4. doi: 10.1016/j.jpeds.2010.07.021. Epub 2010 Sep 17. PMID 20850761
- [Background] Hewett TE, Myer GD, Ford KR. Anterior cruciate ligament injuries in female athletes: Part 1, mechanisms and risk factors. Am J Sports Med. 2006 Feb;34(2):299-311. doi: 10.1177/0363546505284183. PMID 16423913
- [Background] Murphy DF, Connolly DA, Beynnon BD. Risk factors for lower extremity injury: a review of the literature. Br J Sports Med. 2003 Feb;37(1):13-29. doi: 10.1136/bjsm.37.1.13. PMID 12547739
- [Background] Gonzalo-Skok O, Serna J, Rhea MR, Marin PJ. AGE DIFFERENCES IN MEASURES OF FUNCTIONAL MOVEMENT AND PERFORMANCE IN HIGHLY YOUTH BASKETBALL PLAYERS. Int J Sports Phys Ther. 2017 Oct;12(5):812-821. PMID 29181258
- [Background] Tao H, Husher A, Schneider Z, Strand S, Ness B. THE RELATIONSHIP BETWEEN SINGLE LEG BALANCE AND ISOMETRIC ANKLE AND HIP STRENGTH IN A HEALTHY POPULATION. Int J Sports Phys Ther. 2020 Oct;15(5):712-721. doi: 10.26603/ijspt20200712. PMID 33110690
- [Background] Halabchi F, Angoorani H, Mirshahi M, Pourgharib Shahi MH, Mansournia MA. The Prevalence of Selected Intrinsic Risk Factors for Ankle Sprain Among Elite Football and Basketball Players. Asian J Sports Med. 2016 May 23;7(3):e35287. doi: 10.5812/asjsm.35287. eCollection 2016 Sep. PMID 27826402
- [Background] Paz GA, Maia Mde F, Farias D, Santana H, Miranda H, Lima V, Herrington L. KINEMATIC ANALYSIS OF KNEE VALGUS DURING DROP VERTICAL JUMP AND FORWARD STEP-UP IN YOUNG BASKETBALL PLAYERS. Int J Sports Phys Ther. 2016 Apr;11(2):212-9. PMID 27104054
- [Background] Steffen K, Nilstad A, Kristianslund EK, Myklebust G, Bahr R, Krosshaug T. Association between Lower Extremity Muscle Strength and Noncontact ACL Injuries. Med Sci Sports Exerc. 2016 Nov;48(11):2082-2089. doi: 10.1249/MSS.0000000000001014. PMID 27327027
- [Background] Powers CM. The influence of abnormal hip mechanics on knee injury: a biomechanical perspective. J Orthop Sports Phys Ther. 2010 Feb;40(2):42-51. doi: 10.2519/jospt.2010.3337. PMID 20118526
- [Background] Kulas AS, Hortobagyi T, DeVita P. Trunk position modulates anterior cruciate ligament forces and strains during a single-leg squat. Clin Biomech (Bristol). 2012 Jan;27(1):16-21. doi: 10.1016/j.clinbiomech.2011.07.009. Epub 2011 Aug 11. PMID 21839557
- [Background] Biabanimoghadam M, Motealleh A, Cowan SM. Core muscle recruitment pattern during voluntary heel raises is different between patients with patellofemoral pain and healthy individuals. Knee. 2016 Jun;23(3):382-6. doi: 10.1016/j.knee.2016.01.008. Epub 2016 Feb 9. PMID 26873794
- [Background] Kerkhoffs GM, van den Bekerom M, Elders LA, van Beek PA, Hullegie WA, Bloemers GM, de Heus EM, Loogman MC, Rosenbrand KC, Kuipers T, Hoogstraten JW, Dekker R, Ten Duis HJ, van Dijk CN, van Tulder MW, van der Wees PJ, de Bie RA. Diagnosis, treatment and prevention of ankle sprains: an evidence-based clinical guideline. Br J Sports Med. 2012 Sep;46(12):854-60. doi: 10.1136/bjsports-2011-090490. Epub 2012 Apr 20. PMID 22522586
- [Background] Shultz SJ, Schmitz RJ, Benjaminse A, Collins M, Ford K, Kulas AS. ACL Research Retreat VII: An Update on Anterior Cruciate Ligament Injury Risk Factor Identification, Screening, and Prevention. J Athl Train. 2015 Oct;50(10):1076-93. doi: 10.4085/1062-6050-50.10.06. Epub 2015 Sep 4. No abstract available. PMID 26340613
- [Background] Delahunt E, Remus A. Risk Factors for Lateral Ankle Sprains and Chronic Ankle Instability. J Athl Train. 2019 Jun;54(6):611-616. doi: 10.4085/1062-6050-44-18. Epub 2019 Jun 4. PMID 31161942
- [Background] Cowling EJ, Steele JR. Is lower limb muscle synchrony during landing affected by gender? Implications for variations in ACL injury rates. J Electromyogr Kinesiol. 2001 Aug;11(4):263-8. doi: 10.1016/s1050-6411(00)00056-0. PMID 11532597
- [Background] Butler RJ, Crowell HP 3rd, Davis IM. Lower extremity stiffness: implications for performance and injury. Clin Biomech (Bristol). 2003 Jul;18(6):511-7. doi: 10.1016/s0268-0033(03)00071-8. PMID 12828900
- [Background] Podraza JT, White SC. Effect of knee flexion angle on ground reaction forces, knee moments and muscle co-contraction during an impact-like deceleration landing: implications for the non-contact mechanism of ACL injury. Knee. 2010 Aug;17(4):291-5. doi: 10.1016/j.knee.2010.02.013. Epub 2010 Mar 29. PMID 20303276
- [Background] Pollard CD, Sigward SM, Ota S, Langford K, Powers CM. The influence of in-season injury prevention training on lower-extremity kinematics during landing in female soccer players. Clin J Sport Med. 2006 May;16(3):223-7. doi: 10.1097/00042752-200605000-00006. PMID 16778542
- [Background] Fort-Vanmeerhaeghe A, Gual G, Romero-Rodriguez D, Unnitha V. Lower Limb Neuromuscular Asymmetry in Volleyball and Basketball Players. J Hum Kinet. 2016 Apr 13;50:135-143. doi: 10.1515/hukin-2015-0150. eCollection 2016 Apr 1. PMID 28149351